CLINICAL TRIAL: NCT05532956
Title: Evaluation of the Impact of Tricuspid Regurgitation on Patients Lives. Exploration of Experience and Impact on a Daily Basis.
Acronym: EVOQUE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gérond'if (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00641-42
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Severe Tricuspid Regurgitation Medically Treated and Not Operated (Without Valve Replacement or Repair)
Keywords: Severe tricuspid regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individual semi-structured interview: A semi-structured individual interview lasting a maximum of 1.5 hour ,conducted by a psychologist, remotely (telephone, videoconference) or at home
- Collective interview: Group interviews lasting a maximum of 2 hours will consolidate the information obtained during individual interviews

SUMMARY:
The purpose of this study is to objectively assess the impact of the pathology on the patient's life so as to best inform the choices of evaluators "the French National Authority for Health" (HAS) and decision makers "the Economics Committee for Health Products" (CEPS) through the expression of the patients' feelings themselves.

For this, the study will assess the impact of severe tricuspid insufficiency and its symptoms on the quality of life of patients from a physical, psychological and social point of view.

DETAILED DESCRIPTION:
Patients eligible for this study are selected by their cardiologist to participate in one of two interviews:

* Individual semi-structured interview lasting 45 minutes to 1.5 hours conducted by a psychologist These interviews are recorded (voice recording by dictaphone). They address the experience of patients with different degrees of severity of the pathology (severe, massive or torrential regurgitation), questioning the different dimensions of the impact of tricuspid regurgitation on their life, as well as the hierarchy of consequences for their lives and their daily lives.
* Collective interview lasting 1.5 hours to 2 hours which allows to consolidate the information obtained during the individual interviews in order to best assess the impact of the tricuspid regurgitation on the daily life and the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, at least 60 years old,
* Suffering from isolated severe tricuspid insufficiency,
* Symptomatic despite medical treatment,
* Without tricuspid surgery or transcatheter tricuspid surgery, and/or not eligible for surgery,
* Potentially eligible for tricuspid transcatheter therapy (repair or replacement), without considering purely anatomical criteria related to the valve,
* Not suffering from refractory heart failure (stage D) requiring heart transplant or DMCA (mechanical circulatory assist device),
* Without cognitive impairment,
* Not suffering from severe deafness,
* Speaking and understanding French,
* Person not under legal protection and not deprived of liberty

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe tricuspid regurgitation treated medically and not operated (without valve replacement or repair)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of severe tricuspid insufficiency and its symptoms on patients' quality of life | 4 hours
  These are individual interviews conducted by a psychologist and collective support to consolidate the information obtained during the individual interviews.
  This is a purely qualitative analysis. It is not intended to create a new questionnaire or validate existing questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Caroline BACLET-ROUSSEL, Study Chair — Psychologist, Project and Research Manager, Gérond'if